CLINICAL TRIAL: NCT04289805
Title: A Multicenter Prospective coHort Study of Controlled Ovarian Stimulation in Newly Diagnosed Breast Cancer PatiEnts (fAMHOPE)
Brief Title: Controlled Ovarian Stimulation in Newly Diagnosed Breast Cancer PatiEnts (fAMHOPE)
Acronym: fAMHOPE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study had to be terminated due to the new European legislation on drug studies. This legislation requires all studies aimed at evaluating treatments to be registered as such, even in the context of Standard of Care.
Sponsor: Erasme University Hospital (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SRB_201808_163
Record Dates: First submitted 2019-07-17; First posted 2020-02-28 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasm Malignant Female
Keywords: Fertility preservation; Letrozole; Ovarian stimulation
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: 3 groups:
  * 113 patients in the standard-stimulated cohort,
  * 113 patients in the letrozole-stimulated cohort,
  * 339 patients in the non-stimulated cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard-stimulated cohort (Active Comparator): this cohort includes all newly diagnosed breast cancer patients who are candidates to receive (neo)adjuvant chemotherapy and wish to preserve their fertility by undergoing oocyte/embryo cryopreservation at the French participating centres.
  Interventions: Other: standard-stimulated cohort
- letrozole-stimulated cohort (Experimental): this cohort includes all newly diagnosed breast cancer patients who are candidates to receive (neo)adjuvant chemotherapy and wish to preserve their fertility by undergoing oocyte/embryo cryopreservation at the Belgian participating centres.
  Interventions: Drug: Letrozole
- non-stimulated cohort (No Intervention): this cohort includes all newly diagnosed breast cancer patients who are candidates to receive (neo)adjuvant chemotherapy and who have access to the Fertility Clinics in all the participating centres but are not willing to preserve their fertility by undergoing oocyte/embryo cryopreservation.

INTERVENTIONS:
Drug: Letrozole — Patients start ovarian stimulation protocol according to their menstrual cycle phase at enrollment (standard or "random start"). Ovarian stimulation includes gonadotropins administration in a GnRH antagonist protocol.
  "Standard Protocol": letrozole is orally administered (5mg/d) from cycle day 2-3 throughout the ovarian stimulation with gonadotropins protocol until ovulation triggering.
  "Random start" protocol: letrozole is administered throughout the stimulation together with gonadotropins.
  GnRH antagonist is administered at cycle day 7 or as soon as at least one follicle reaches 12-14 mm.
  Oocytes are collected 36h after ovulation triggering with GnRH agonist.
  Other Names: Controlled Ovarian Stimulation (COS)
  Arms: letrozole-stimulated cohort
Other: standard-stimulated cohort — Patients start ovarian stimulation protocol according to their menstrual cycle phase at enrollment (standard or "random start"). Ovarian stimulation includes gonadotropins administration in a GnRH antagonist protocol.
  "Standard Protocol": Gonadotrophins started from cycle day 2-3 throughout the ovarian stimulation until ovulation triggering.
  "Random start" protocol: Gonadotrophins started at any time of the cycle and throughout the stimulation.
  GnRH antagonist is administered at cycle day 7 or as soon as at least one follicle reaches 12-14 mm.
  Oocytes are collected 36h after ovulation triggering with GnRH agonist.
  Other Names: COS
  Arms: standard-stimulated cohort

SUMMARY:
This is a multicenter hospital-based prospective cohort study conducted in institutions with known expertise in performing oocytes/embryo freezing for fertility preservation. The study aims at refining the understanding of the efficacy and safety of controlled ovarian stimulation with or without letrozole in young women with newly diagnosed breast cancer who are candidates to receive (neo)adjuvant chemotherapy.

DETAILED DESCRIPTION:
Patients enrolled in this study undergo standard or "random start" ovarian stimulation with Gonadotropins using antagonist protocol before the beginning of chemotherapy. Ovulation is triggered in all patients with a Gonadotropin Releasing Hormone-GnRH agonist.

After retrieval, oocytes are denuded and matured oocytes are subjected to fertilization before embryo freezing or direct vitrification.

Primary objective is to evaluate the efficacy of performing a controlled ovarian stimulation with or without letrozole in young women with newly diagnosed breast cancer who are candidates to receive (neo)adjuvant chemotherapy in terms of mature oocytes collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive non-metastatic breast cancer (i.e. stage I to III);
* Breast cancer diagnosis ≥18 and ≤ 40 years;
* No prior history of gonadotoxic treatments;
* Fertility preservation counseling for fertility preservation;
* Written inform consent;
* FSH < 20 UI/L and/or antra-follicular count ≥ 6 (follicles of 2-9 mm) and/or AMH ≥ 6 pmol (only applicable for patients who undergo controlled ovarian stimulation for embryo/oocyte cryopreservation).

Exclusion Criteria:

* Newly diagnosed stage IV breast cancer (i.e. de novo metastatic breast cancer);
* Prior diagnosis of other malignancies before breast cancer.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of the ovarian stimulation and oocyte collection procedure: Number of mature oocytes collected | an average of 2 weeks after inclusion
  Number of mature oocytes collected

SECONDARY OUTCOMES:
Number of patient with adverse events due to COS: OHSS | Through treatment procedure, an average of 2 weeks after inclusion
  Adverse events reporting during COS (Ovarian Hyperstimulation syndrome-OHSS)
Characteristics of Ovarian stimulation: total gonadotropin doses | An average of 2 weeks after inclusion
  Total gonadotropin doses (International Unit- IU)
Characteristics of Ovarian stimulation: duration of the COS | An average of 2 weeks after inclusion
  duration of the COS (days)
Characteristics of Ovarian stimulation: type of stimulation | An average of 2 weeks after inclusion
  type of stimulation (standard or random-start).
Efficacy of the ovarian stimulation and oocyte collection: Maturation rate | An average of 2 weeks after inclusion
  Maturation rate (number of total oocyte collected/number of mature oocytes)
Outcomes of assisted reproductive technology procedures | Through study completion, 5 years
  Number of pregnancies and outcomes (premature delivery, miscarriage, abortion, delivery healthy babies, congenital malformation).
Anticancer therapies effect on ovarian function: progesterone | Inclusion, an average of 2 weeks, 6 months, 18 months, 30 months, 60 months
  Hormonal measurements Progesterone ng/ml
Anticancer therapies effect on ovarian function: AMH | Inclusion, an average of 2 weeks, 6 months, 18 months, 30 months, 60 months
  Anti-Mullerian Hormone (AMH) measurements AMH ng/ml
Anticancer therapies effect on ovarian function: FSH | Inclusion, an average of 2 weeks, 6 months, 18 months, 30 months, 60 months
  Follicle-Stimulating Hormone (FSH) measurements FSH IU/L
Anticancer therapies effect on ovarian function: E2 | Inclusion, an average of 2 weeks, 6 months, 18 months, 30 months, 60 months
  Hormonal measurements E2 pg/ml
Anticancer therapies effect on ovarian function | An average 18 months, 30 months, 60 months after inclusion
  Amenorrhea rate (6months without spontaneous menstruation)
Oncological outcomes 1 | 5 years
  Invasive disease-free survival (iDFS)
Oncological outcomes 2 | 5 years
  breast cancer-free interval (BCFI)
Oncological outcomes 3 | 5 years
  overall survival (OS)
Circulating breast cancer cells level before stimulation | Inclusion
  circulating tumor DNA (ctDNA)
Circulating breast cancer cells level after stimulation | average of 2weeks after inclusion
  circulating tumor DNA (ctDNA)
Number of patient with adverse events due to egg collection | An average of 2 weeks after inclusion
  bleeding
Number of patient with adverse events due to egg collection | An average of 2 weeks after inclusion
  pelvic infection
Efficacy of the in vitro fertilization procedure: Fertilization rate | Through study completion, 5 years
  Fertilization rate (number of oocyte fertilized/number of embryo obtained)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Demeestere, MD, PhD, Study Director — CUB-Hôpital Erasme; Matteo Lambertini, MD, PhD, Study Chair — ULB; Christine Decanter, MD, Study Chair — CHRU LILLE
Locations (6):
- Belgium (3):
  - CUB-Hôpital Erasme, Brussels
  - CHIREC- Hospital Delta, Brussels
  - CHC-Saint Vincent, Liège
- France (2):
  - Centre Oscar Lambret, Lille
  - CHRU Lille, Lille
- Ospedale San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT04289805/Prot_SAP_000.pdf